CLINICAL TRIAL: NCT02446210
Title: Targeted Neuroplasticity After Spinal Cord Injury
Brief Title: Neuroplasticity After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Monica Perez, Chair Arms + Hands Lab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STU0020971; R01NS076589-01 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-05-18 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injury
Keywords: SCI; Neural Control; Bilateral Movement; TMS
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Controls Group (Active Comparator): Magstim 200 magnetic stimulator for Transcranial Magnetic Stimulation and Peripheral Nerve Stimulation
  Interventions: Device: Magstim 200; Device: Digitimer electrical stimulator
- Spinal Cord Injury Group (Active Comparator): Magstim 200 magnetic stimulator for Transcranial Magnetic Stimulation and Peripheral Nerve Stimulation
  Interventions: Device: Magstim 200; Device: Digitimer electrical stimulator

INTERVENTIONS:
Device: Magstim 200 — Transcranial Magnetic Stimulation
Device: Digitimer electrical stimulator — Transcranial Magnetic Stimulation paired with Electrical Peripheral Nerve Stimulation
  Other Names: Electrical stimulation

SUMMARY:
The long-term goal is to acquire scientific knowledge that can be used to develop mechanistic-driven intervention strategies aiming at restoring upper and lower-limb motor function in individuals with cervical or thoracic spinal cord injury (SCI). The proposed project will examine cortical, corticospinal, and spinal contribution to bilateral hand and arm muscle activity during bilateral movements and spinal contributions to lower limb muscle activity. By comparing changes in different sites within the Central Nervous System (CNS), the investigators may also identify key mechanisms that might be differentially affected by the injury, plasticity, and training.

DETAILED DESCRIPTION:
If the participant qualifies to take part in this research study, they will be asked to participate in 15-190 study visits,to complete the experimental procedures. These procedures have been broken up into "Phases" and will be completed in any order. Phase I and Phase IIa includes 2-30 total visits - approximately 2-3 hours each to measure arm and finger strength and ability to move. Phase IIb includes 2-30 total visits - approximately 2-3 hours each, to measure leg strength and ability to move. Phase IIIa includes up to 40 total visits - approximately 2 hours each, the investigator will again evaluate the participant's ability to use both arms. The participant will be asked to complete a series of tasks such as stacking checkers, turning over cards, squeeze a device to determine how strong their grip is, and see how well they are able to feel sensations on the surface of their skin. The investigators will complete these assessments at pre-determined times during the study participation. Phase IIIb includes up to 40 total visits - approximately 2 hours each, the investigator will again evaluate the participant's ability to use both legs. Assessments of the participant's legs will include walking around the lab space, how well they can bend their ankles and hips, and how well they are able to feel sensations on the surface of the participant's skin.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for individuals with SCI:

  * Male and females between ages 18-85 years
  * SCI (≥1 month after injury)
  * Cervical, thoracic or lumbar injury above L2 (tetraplegia)Intact (level 2) or impaired (level 1) but not absent (level 0) lower motor neuron innervations in dermatomes C6, C7 and C8 during light touch and pin prick stimulus using the American Spinal Injury Association (ASIA) sensory scores (12)
  * The ability to produce a visible precision grip force with both hands
  * Individuals who have the ability to pick up a small object (large paperclip) from a table independently
  * Ability to perform 30° or more of elbow flexion and extension.
  * The ability to perform a visible contraction with dorsiflexor and hip flexor muscles
  * The ability to ambulate a few steps with or without an assistive device

Inclusion criteria for healthy controls:

* Male and females between ages 18-85 years
* Right handed
* Able to complete precision grips with both hands
* Able to complete full elbow flexion-extension with both arms.
* Able to walk and complete lower-limb tests with both legs.

Exclusion Criteria:

* Exclusion criteria for individuals with SCI and Healthy Controls:

  * Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
  * Any debilitating disease prior to the SCI that caused exercise intolerance
  * Premorbid, ongoing major depression or psychosis, altered cognitive status
  * History of head injury or stroke
  * Pacemaker
  * Metal plate in skull
  * History of seizures
  * Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants
  * Pregnant females
  * Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida or herniated cervical disk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-01-27 (Estimated); Study Completion 2023-01-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reduced motor cortical excitability | 5 months
  Measured by Electroencephalogram/Electromyography and Electromyography/Electromyography coherence

SECONDARY OUTCOMES:
Number of participants with enhance voluntary motor output in upper limbs | 5 months
  Measured by spike-timing-dependent plasticity
Number of participants with enhance voluntary motor output in lower limbs | 5 months
  Measured by spike-timing-dependent plasticity

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PhD, PT, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States